CLINICAL TRIAL: NCT01197196
Title: Behavioral Weight Loss as a Treatment for Migraine in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0068-10; R01NS077925-01A1 (NIH)
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2016-09

CONDITIONS: Migraine; Obesity
Keywords: Migraine; Obesity; Weight loss; Lifestyle; Behavior
MeSH Terms: conditions — Migraine Disorders; Obesity; Weight Loss; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral weight loss (Experimental)
  Interventions: Behavioral: Behavioral Weight Loss Intervention
- Migraine Education (Active Comparator)
  Interventions: Other: Migraine Education

INTERVENTIONS:
Behavioral: Behavioral Weight Loss Intervention — Participants assigned to this condition will receive an intensive group-based lifestyle program modeled after the DPP and Look AHEAD trials. Participants will attend 16 weekly sessions involving provision of behavioral goals and strategies to modify diet and exercise behaviors in order to achieve a weight loss of at least 7% of initial body weight.
  Arms: Behavioral weight loss
Other: Migraine Education — Participants assigned to this condition (Healthy Living for Migraine Relief [HLMR]) will receive basic education and didactic instruction in migraine headaches and treatments that are the standard of care. Participants will attend 4 months of weekly group lectures focused on 3 different major topic areas: 1) migraine symptomatology and pathophysiology, 2) standard abortive and preventive pharmacological treatment options, and 3) standard and alternative non-pharmacological treatment options.
  Arms: Migraine Education

SUMMARY:
This study involves a randomized controlled trial to test the efficacy of behavioral weight loss as a treatment for migraine in obese females aged 18 to 50 years. The primary aim is to examine whether participants assigned to a behavioral weight loss treatment condition report greater pre- to post-treatment reductions in migraine headache frequency than participants assigned to a migraine education condition.

DETAILED DESCRIPTION:
Migraine is a highly prevalent, debilitating and costly disorder. Eighteen percent of women and 6% of men are affected by migraine; a neurovascular disorder characterized by severe recurrent headache pain episodes involving nausea, photophobia, phonophobia and aversion to physical activity.

There is increasing evidence that obesity exacerbates migraine. Obesity is associated with more frequent headaches in episodic migraineurs, and is a risk factor for progression to chronic migraine. Several plausible mechanisms have been proposed to underlie the migraine-obesity link including common pro-inflammatory processes, psychological conditions that are comorbid to both disorders (e.g., depression), and similar behavioral risk factors (e.g., low physical activity and high fat intake).

No research to date has examined the impact of standard behavioral weight loss programs on migraine in obese adults. Behavioral weight loss programs focused on improving diet and physical activity consistently produce weight losses of 8-10 kg at 6 months which reduces the risk of diabetes and improves cardiovascular disease risk factors. Weight loss may also improve each of the physiological, psychological, and behavioral pathways that purportedly link migraine and obesity. Thus, behavioral weight loss programs may serve as an innovative approach to treating migraine headaches.

This study involves a randomized controlled trial to examine the efficacy of behavioral weight loss as a treatment for migraine. One hundred and forty obese females who meet research criteria for migraine, as confirmed by a study neurologist and completion of an electronic headache diary will be assigned to 16 weekly group sessions of either: (1) Behavioral weight loss (BWL) treatment (n=70) or (2) Healthy Living for Migraine Relief (HLMR) education (n=70). BWL will provide a combination of empirically validated diet and exercise prescriptions and behavior change strategies such as self-monitoring, goal-setting and stimulus control. HLMR will provide education on migraine and pharmacological and behavioral (e.g., stress management) treatments. Both groups will use smartphones to record their headaches for 4 weeks at a time during pre-treatment, post-treatment, and the end of a 16-week weight maintenance period. Weight and other potential physiological (inflammation), psychological (depression), and behavioral (diet and physical activity) mediators of the treatment effect will be assessed at the end of treatment for tests of prospective effects on migraine days at post-treatment. The primary hypothesis is that BWL participants will report greater pre- to post-treatment reductions in number of migraine days than HLMR participants.

ELIGIBILITY:
Inclusion criteria:

* Neurologist-confirmed diagnosis of migraine with or without aura
* Experience at least 3 headaches and 4-20 headache days per month
* Body Mass Index of 25.0-49.9 kg/m2

Exclusion criteria:

* Have primary headache disorder other than migraine or tension-type headache
* Have both migraine and tension-type headache and are unable to distinguish the two headache types and/or report 2 or more tension-type headaches per month
* Have a secondary headache disorder
* Have initiated or changed prophylactic medications within 2 months of study entry, or intend to change these medications during the trial
* Have changed medications used to abort migraine attacks, treat depression, or provide oral contraception within 2 months of study entry, or intend to change these medications during the trial.
* Have experienced recent weight loss (>=5% within the past 6 months), are currently involved in a commercial weight loss program, are presently taking weight loss medications, or have had bariatric surgery.
* Are pregnant, were pregnant within the last 6 months, or plan to become pregnant during the trial.
* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire. Individuals reporting joint problems, prescription medication usage, or other medical conditions that could limit exercise participation will be required to obtain written physician consent to participate.
* Have been diagnosed with cancer or are currently undergoing cancer treatment.
* Are unable to read or understand the study materials.
* Report any condition that in the opinion of investigators would reduce the likelihood of adherence to the headache monitoring protocol or clinical trial prescriptions, including terminal illness, planning to relocate, or a history of substance abuse, bulimia nervosa, or other significant psychiatric problems.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2012-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in the number of migraine headache days | Baseline, end of treatment, end of 16-week weight maintenance period
  Measured via 28-day mobile smartphone headache diary

SECONDARY OUTCOMES:
Change in body weight | baseline, end of treatment, end of 16-week weight maintenance period
Changes in serum inflammatory markers (C-reactive protein, Interleukin-6) | Baseline, end of treatment
  Changes in inflammation will be tested as a mediator of the treatment effect.
Changes in depression | Baseline, end of treatment
  Changes in depressive symptoms will be tested as a mediator of the treatment effect.
Changes in physical activity | Baseline, end of treatment
  Physical activity will be objectively assessed via a multi-sensor monitor. Changes in physical activity will be tested as a mediator of the treatment effect.
Changes in fat intake and other diet/eating behavior components | Baseline, end of treatment
  Diet and eating behavior will be measured via a multi-call 24 hour dietary recall procedure. Changes in fat intake will be tested as as mediator of the treatment effect.

OTHER OUTCOMES:
Changes in additional migraine headache parameters | Baseline, end of treatment
  Additional headache parameters include daily headache activity (severity and duration of attacks, clinical features (photophobia, phonophobia, nausea), abortive medication usage, allodynia, and headache management self-efficacy.
Changes in waist circumference and cardiometabolic risk factors | Baseline, end of treatment
  Cardiometabolic risk factors will include systolic and diastolic blood pressure, total and HDL cholesterol, triglycerides, and insulin sensitivity.
Changes in anxiety symptoms and level of psychological stress. | Baseline, end of treatment
Changes in sleep quality | Baseline, end of treatment
  Sleep duration and quality will be assessed via self-report and objectively using a multi-sensor monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Dale S. Bond, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Smith KE, Thomas JG, Steffen KJ, Lipton RB, Farris SG, Pavlovic JM, Bond DS. Naturalistic assessment of patterns and predictors of acute headache medication use among women with comorbid migraine and overweight or obesity. Transl Behav Med. 2021 Aug 13;11(8):1495-1506. doi: 10.1093/tbm/ibab027. PMID 33823051
- [Derived] Farris SG, Thomas JG, Kibbey MM, Pavlovic JM, Steffen KJ, Bond DS. Treatment effects on pain catastrophizing and cutaneous allodynia symptoms in women with migraine and overweight/obesity. Health Psychol. 2020 Oct;39(10):927-933. doi: 10.1037/hea0000920. Epub 2020 Jul 13. PMID 32658497
- [Derived] Lillis J, Thomas JG, Lipton RB, Rathier L, Roth J, Pavlovic J, O'Leary KC, Bond DS. The Association of Changes in Pain Acceptance and Headache-Related Disability. Ann Behav Med. 2019 Jun 4;53(7):686-690. doi: 10.1093/abm/kay076. PMID 30289426
- [Derived] Farris SG, Thomas JG, Abrantes AM, Lipton RB, Pavlovic J, Smitherman TA, Irby MB, Penzien DB, Roth J, O'Leary KC, Bond DS. Pain worsening with physical activity during migraine attacks in women with overweight/obesity: A prospective evaluation of frequency, consistency, and correlates. Cephalalgia. 2018 Oct;38(11):1707-1715. doi: 10.1177/0333102417747231. Epub 2017 Dec 13. PMID 29237284
- [Derived] Bond DS, Thomas JG, Lipton RB, Roth J, Pavlovic JM, Rathier L, O'Leary KC, Evans EW, Wing RR. Behavioral Weight Loss Intervention for Migraine: A Randomized Controlled Trial. Obesity (Silver Spring). 2018 Jan;26(1):81-87. doi: 10.1002/oby.22069. Epub 2017 Nov 27. PMID 29178659
- [Derived] Bond DS, Buse DC, Lipton RB, Thomas JG, Rathier L, Roth J, Pavlovic JM, Evans EW, Wing RR. Clinical Pain Catastrophizing in Women With Migraine and Obesity. Headache. 2015 Jul-Aug;55(7):923-33. doi: 10.1111/head.12597. Epub 2015 Jun 18. PMID 26087348
- [Derived] Bond DS, Thomas JG, O'Leary KC, Lipton RB, Peterlin BL, Roth J, Rathier L, Wing RR. Objectively measured physical activity in obese women with and without migraine. Cephalalgia. 2015 Sep;35(10):886-93. doi: 10.1177/0333102414562970. Epub 2014 Dec 4. PMID 25475207
- See also: Related Info — http://www.weightresearch.org/fundedgrants.html